CLINICAL TRIAL: NCT03818789
Title: Mindfulness and Acceptance for Exercise in Anxiety
Brief Title: Acceptance and Mindfulness for Exercise in Anxiety
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Emily Carl, Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016-11-0091
Record Dates: First submitted 2018-10-31; First posted 2019-01-28 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): A mindfulness training is applied to see if it supports exercise endurance in-lab and during follow-up
  Interventions: Behavioral: Mindfulness and acceptance training
- Control (Placebo Comparator): A study skills video is shown intended to have no effect on exercise but to match for time.
  Interventions: Behavioral: Study skills video

INTERVENTIONS:
Behavioral: Mindfulness and acceptance training — A breathing mediation, body scan, talking about acceptance, and presence activity are used. All are low-impact and expected to cause no distress
  Arms: Mindfulness
Behavioral: Study skills video — A YouTube video describing study skills and suggested habits is used as a control condition.
  Arms: Control

SUMMARY:
Anxiety is a common experience, with the U.S. lifetime prevalence of any anxiety disorder at 28.8%. Exercise has shown large effect sizes relative to controls in reducing mood and anxiety symptoms. An anxious population generally has more difficulty when beginning or increasing an exercise regimen, due to a higher level of sensitivity to discomfort. Mindfulness practices may be helpful in improving adherence to an exercise program. A similar study has shown that mindfulness may reduce perceived effort and make exercise more enjoyable. Furthermore, mindfulness has been shown to be an effective intervention in reducing anxiety and physical discomfort. The investigators intend to use a brief intervention incorporating strategies of mindfulness and Acceptance and Commitment Therapy (ACT) in conjunction with exercise to ease the transition into regular/increased physical exercise. Measures of anxiety sensitivity and perceived stress will be included to measure whether they change, and their possible effect as moderating variables on exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

* Students who are enrolled in Psychology 301 at the University of Texas at Austin, as well as adult and student volunteers recruited from the University of Texas at Austin campus and the greater Austin community, who are 18-65 will be eligible for this study.
* Participants must exercise less than 150 minutes per week doing moderate-intensity exercise consistently within the last two months.
* They will have at least mild anxiety, as measured with either a minimum score of 8 on the Beck Anxiety Inventory, or 5 on the Generalized Anxiety Disorder-7.

Exclusion Criteria:

* Those that are at moderate or high risk based on the pre-participation exercise health screening by the American College of Sports Medicine, or any participants that have been advised to not participate in exercise or aerobic activity by a qualified medical provider.
* Those with cardiovascular or pulmonary diseases, immunological diseases, neurological disorders, or have serious bone or joint problems.
* The Beck Depression Inventory's item on suicidality will be actively checked for a response of 2 or 3, with further screening given to those participants using questions from the C-SSRS to screen for current suicidal ideation and past suicidal behavior. Participants who endorse imminent intent or a plan to act on suicidal thoughts will be immediately referred to one of the IMHR's psychologists, or 911 will be contacted if they are at immediate risk of suicidal self-harm. Participants endorsing intent or a specific plan will not be included in the study. Participants expressing suicidal thoughts without imminent intent or a specific plan will be given resources to pursue mental health treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Amount of time run in minutes | During lab visit (day 1 of participation)
  The voluntary decision when to stop exercising on the treadmill in the lab
Amount of time in minutes of vigorous and moderate exercise in following week | One week follow-up
  Amount exercised as assessed by International Physical Activity Questionnaire at follow-up

SECONDARY OUTCOMES:
Anxiety symptoms: Generalized Anxiety Disorder - 7 Scale, Beck Anxiety Inventory | One week follow-up
  These self-report questionnaires assess general anxiety symptoms
Depression symptoms: Beck Depression Inventory | One week follow-up
  This self-report questionnaire assesses depression symptoms
Mindfulness during exercise: State Mindfulness Scale for Physical Activity | Assessed in the lab (day 1 of participation) and at follow-ups one week later
  This self-report questionnaire is designed to assess mindful state specifically during exercise

CONTACTS AND LOCATIONS:
Locations (1):
- College of Liberal Arts, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided